CLINICAL TRIAL: NCT02499913
Title: Contingency Management to Reduce Alcohol Use in a Soup Kitchen Sample
Acronym: SK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Carla Rash, Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-177-1; P60AA003510 (NIH)
Record Dates: First submitted 2015-07-14; First posted 2015-07-16 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Alcohol Abuse; Contingency Management
MeSH Terms: conditions — Alcoholism | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- breath alcohol monitoring (Active Comparator): Breath alcohol samples and self-reports of drinking will be collected once daily at lunch and will be used as objective indicators of recent alcohol use.
  Interventions: Behavioral: breath alcohol monitoring
- breath monitoring plus prize contingency management (Experimental): Breath alcohol samples and self-reports of drinking will be collected once daily at lunch and will be used as objective indicators of recent alcohol use. Participants of this group earn opportunities to draw cards from a prize bowl for negative breath samples.
  Interventions: Behavioral: breath alcohol monitoring; Behavioral: contingency management

INTERVENTIONS:
Behavioral: breath alcohol monitoring — Daily breath alcohol monitoring
Behavioral: contingency management — Participants can earn chance to win prizes for negative breath alcohol samples.
  Arms: breath monitoring plus prize contingency management

SUMMARY:
Alcohol use and alcohol-related disorders are highly prevalent in soup kitchen users, and this population is overrepresented by minorities and disproportionately affected by alcohol-related morbidity and mortality. Contingency management is a behavioral intervention effective in reducing substance use, but few studies have evaluated the efficacy of contingency management in the context of soup kitchens or homeless programs. The investigators found that contingency management, using a twice weekly testing and reinforcement schedule, had benefits for decreasing drinking in individuals receiving services at a homeless shelter. This study will replicate and extend these earlier findings to a soup kitchen population using more sophisticated alcohol monitoring procedures to better assess the extent of drinking in this group and in response to a contingency management intervention reinforcing submission of negative breath samples. Specifically, 40 hazardous drinkers recruited from a soup kitchen will be randomly assigned to one of two conditions: alcohol monitoring or the same plus reinforcement for provision of daily negative breath alcohol samples. The interventions will be in effect for 3 weeks, and all participants will also wear transdermal continuous alcohol monitors during the intervention period. Objective and subjective indices of alcohol consumption will be evaluated and compared between and within the treatment conditions. This pilot project will provide information regarding the effect size of contingency management reinforcing negative breath samples in an important health disparities group, and results from this study will guide subsequent grant applications focusing on methods to decrease drinking in this underserved population.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18
* frequent soup kitchen users who drink alcohol
* willing to wear transdermal alcohol monitor for 3 weeks
* willing to sign a property transfer form and return SCRAMx equipment

Exclusion Criteria:

* uncontrolled, severe psychopathology and/or severe cognitive impairment
* non-English speaking
* in recovery for pathological gambling
* has a medical condition that would interfere with transdermal alcohol readings
* legal charges pending that are likely to lead to incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
efficacy of contingency management relative to monitoring only | week 4
  longest duration of abstinence

CONTACTS AND LOCATIONS:
Overall Officials: Carla Rash, Ph.D., Principal Investigator — UConn Health
Locations (1):
- Friendship Center, New Britain, Connecticut, United States